CLINICAL TRIAL: NCT06449339
Title: Baveno VII Criteria-guided Initiation of Non-selective Beta Blocker in Patients With Compensated Advanced Chronic Liver Disease to Reduce Hepatic Decompensation: an Open-label Randomised Controlled Trial
Brief Title: Non-selective Beta-blocker in Compensated Advanced Chronic Liver Disease
Acronym: BB_cACLD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Singapore General Hospital (Other); University of Palermo (Other); University of Malaya (Other); Shanghai Jiao Tong University School of Medicine (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Principal Investigator, Jimmy Che-To Lai, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.521-T
Record Dates: First submitted 2024-05-29; First posted 2024-06-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Portal Hypertension; Hepatic Decompensation; Advanced Chronic Liver Disease
Keywords: compensated advanced chronic liver disease; non-selective beta-blocker; Baveno VII; hepatic decompensation
MeSH Terms: conditions — Hypertension, Portal | interventions — Carvedilol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-selective beta-blocker (NSBB) (Experimental): oral carvedilol 6.25mg-50mg daily
  Interventions: Drug: Carvedilol
- Conventional (No Intervention): Not on oral carvedilol

INTERVENTIONS:
Drug: Carvedilol — Patients in the NSBB arm will receive generic carvedilol. The starting dose of oral carvedilol is 6.25mg daily (to be taken once or twice per day) and can be adjusted at each scheduled visit (either by increasing the dosage or frequency of dose administration) according to patients' tolerance, as well as the blood pressure and pulse rate that the systolic blood pressure should be not lower than 90 mmHg and pulse rate not lower than 55 beats per minute. The dosage of carvedilol can also be titrated or discontinued at unscheduled visit according to patient's condition. In case carvedilol is discontinued, it can be resumed from the starting dose at next scheduled visit if there is no contraindication for carvedilol. The dose of carvedilol will be kept at 6.25-12.5mg per day unless there are additional non-hepatic indications such as arterial hypertension or cardiac disease warranting higher carvedilol dosage. The maximum allowed dose of carvedilol is 50mg daily as per drug instruction.
  Arms: non-selective beta-blocker (NSBB)

SUMMARY:
The goal of this randomised controlled trial is to evaluate the effect of carvedilol (a non-selective beta-blocker) in patients with compensated advanced chronic liver disease under clinically significant portal hypertension or the grey zone of Baveno VII criteria.

The main question it aims to answer is:

Does carvedilol reduce hepatic decompensation and mortality in these patients despite the absence of varices needing treatment.

Researchers will compare carvedilol to no carvedilol to see if carvedilol can prevent hepatic decompensation and mortality.

Participants will either take carvedilol or not taking carvedilol for 5 years with regular clinic visit for checkups and investigations, including blood tests, ultrasonography of the liver, upper gastrointestinal endoscopy, transient elastography.

DETAILED DESCRIPTION:
The study is a multi-centre, open-label, randomised controlled trial conducted in Prince of Wales Hospital, a tertiary academic hospital in Hong Kong, as well as other international study sites. Eligible patients will be randomised to NSBB arm (i.e. receiving carvedilol) or conventional arm (i.e. not receiving carvedilol), aiming to test the hypothesis that Baveno VII criteria-guided carvedilol treatment in compensated advanced chronic liver disease (cACLD) patients in grey zone or with clinically significant portal hypertension (CSPH) is superior to not treating them in the absence of high-risk varices (HRV), in terms of prevention of first occurrence of hepatic decompensation and mortality. Consecutive patients in the participating study sites with cACLD fulfilling the high-risk grey zone and CSPH criteria by LSM and platelet count will be invited to this study. The patients will undergo oesophagogastroduodenoscopy (OGD) for screening of oesophageal varices (OV). Those without HRV will be randomised into NSBB and conventional arms. Patients in the NSBB arm will be started on carvedilol. Those in the conventional arm will not receive NSBB as per current standard of practice. The expected accrual duration is 24 months with an interim analysis to be performed when all enrolled patients have reached 1 year of follow-up or the primary endpoint. The total follow-up duration is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of above
* Established diagnosis of chronic liver disease(s) of the following etiologies

  * Alcohol-related liver disease (ARLD)
  * Chronic hepatitis B (CHB)
  * Chronic hepatitis C (CHC)
  * Metabolic dysfunction-associated steatotic liver disease (MASLD) § Non-obese (BMI <30kg/m2) and obese (BMI ≥30 kg/m2)
* In high-risk grey zone or CSPH, by Baveno VII criteria (for ARLD, CHB, CHC and non-obese MASLD) or ANTICIPATE-NASH model (for obese MASLD) within 6 months from screening

  * Baveno VII criteria (for ARLD, CHB, CHC and non-obese MASLD)

    * LSM ≥25 kPa (CSPH)
    * LSM ≥20 kPa - <25 kPa and platelet count <150 x 10^9/L; or LSM ≥15 kPa - <20 kPa and platelet count <110 x 10^9/L (high-risk grey zone)
  * ANTICIPATE-NASH model (for obese MASLD)

    * Predictive probability for CSPH >90% (CSPH)
    * Predictive probability for CSPH ≥60% - <90% (high-risk grey zone)

Exclusion Criteria:

* Presence of high-risk varices (HRV) (i.e. moderate to large oesophageal varices [OV] or OV with red wale sign) found in OGD
* Current use of non-selective beta-blocker (NSBB) or any use of NSBB within 6 months before

  * Use of selective beta blocker, such as atenolol or metoprolol, is not excluded
  * Selective beta-blocker will be switched to carvedilol in NSBB arm, and will be kept unchanged in conventional arm if there is clinical need for the selective beta-blocker
* Contraindication to NSBB (e.g. Type II/III heart block or baseline bradycardia <60/minute, hypotension with systolic blood pressure (SBP) <100 mmHg, asthma, poorly controlled chronic obstructive pulmonary disease, and peripheral vascular disease)
* Current use of nitrated drugs or any use of nitrated drugs within 6 months before

  o Use of sublingual nitrate, such as glyceryl trinitrate, is not excluded
* Contraindication to OGD (e.g. Intestinal perforation or obstruction)
* Current or history of decompensated liver cirrhosis (i.e. Child's C cirrhosis, prior decompensating events such as ascites, variceal bleeding, hepatic encephalopathy and hepatorenal syndrome)

  o Child's B cirrhosis without decompensating events is not excluded
* Current or history of hepatocellular carcinoma (HCC)
* Current or history of portal vein thrombosis
* Transjugular intrahepatic portosystemic shunt (TIPS)
* Liver transplantation
* Serious medical illness with limited life expectancy of less than 6 months
* Pregnancy
* Unable to obtain or refusal of informed consent from patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2031-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
composite of incident high-risk varices (HRV), hepatic decompensation or death | 5 years
  HRV is defined by moderate to large oesophageal varices (OV) or OV with red wale sign. Hepatic decompensation is defined by the presence of ascites, variceal bleeding or overt hepatic encephalopathy

SECONDARY OUTCOMES:
Number of participants with development of each hepatic decompensation event | 5 years
  Hepatic decompensation events include ascites, variceal bleeding and overt hepatic encephalopathy
Number of participants with development of hepatocellular carcinoma | 5 years
  Development of hepatocellular carcinoma
Change in hepatic function in terms of Child-Pugh score | 5 years
  Higher Child-Pugh score indicates poorer liver condition, vice versa
Change in hepatic function in terms of model for end-stage liver disease (MELD) score | 5 years
  Higher MELD score indicates poorer liver condition, vice versa
Change in liver stiffness measurement (LSM) and spleen stiffness measurement (SSM) | 5 years
  Change in liver and spleen stiffness measurements on transient elastography
Adverse events | 5 years
  Any adverse events during the study period
Number of participants who survive until the last clinic visit | 5 years
  Survival until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Che-To Lai, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the first publication until 15 years after the end of the study
Access Criteria: By email communication

REFERENCES:
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Pons M, Augustin S, Scheiner B, Guillaume M, Rosselli M, Rodrigues SG, Stefanescu H, Ma MM, Mandorfer M, Mergeay-Fabre M, Procopet B, Schwabl P, Ferlitsch A, Semmler G, Berzigotti A, Tsochatzis E, Bureau C, Reiberger T, Bosch J, Abraldes JG, Genesca J. Noninvasive Diagnosis of Portal Hypertension in Patients With Compensated Advanced Chronic Liver Disease. Am J Gastroenterol. 2021 Apr;116(4):723-732. doi: 10.14309/ajg.0000000000000994. PMID 33982942

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT06449339/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT06449339/ICF_001.pdf